CLINICAL TRIAL: NCT02255266
Title: Long-Term Effectiveness of Liraglutide for Treatment of Type 2 Diabetes in Daily Practice
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-4118; U1111-1143-9842 (Other: WHO)
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — No treatment given.

SUMMARY:
This study is conducted in Europe. The aim of this study is to investigate Long-Term Effectiveness of Liraglutide for Treatment of Type 2 Diabetes in daily Practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of age above 18 years as per Victoza® SmPC par.4.2 and 5.1 diagnosed with type 2 diabetes receiving the first prescription of liraglutide in 2011

Exclusion Criteria:

* None. Available data from all eligible patients for each center, will be included

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive subjects initiating liraglutide in 2011 according to Victoza® SmPC meeting the inclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1788 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2015-11-16 (Actual)

PRIMARY OUTCOMES:
Frequency of patients achieving HbA1c reduction of at least 1%-point | Week 0, week 52

SECONDARY OUTCOMES:
Change in HbA1c (Glycosylated haemoglobin)) | Week 0, week 104
Change in body weight | Week 0, week 104
Frequency of patients achieving HbA1c reduction of at least 1%-point | After 4 and 24 months of treatment
Frequency of patients achieving HbA1c target (<=7%) | After 4, 12 and 24 months
Frequency of patients achieving a body weight reduction of at least 3% | After 4, 12 and 24 months
Frequency of patients achieving the composite endpoint consisting in: HbA1c reduction of at least 1%-point and body weight reduction of at least 3% | After 4, 12 and 24 months
Percentage of treatment discontinuation for any reason | At 4, 12 and 24 months
Changes in blood pressure and lipid profile | Week 0, week 104

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Rome, Italy

REFERENCES:
- [Result] Lapolla A, Berra C, Boemi M, Bossi AC, Candido R, Di Cianni G, Frontoni S, Genovese S, Ponzani P, Provenzano V, Russo GT, Sciangula L, Simioni N, Bette C, Nicolucci A; NN2211-4118 Study Group. Long-Term Effectiveness of Liraglutide for Treatment of Type 2 Diabetes in a Real-Life Setting: A 24-Month, Multicenter, Non-interventional, Retrospective Study. Adv Ther. 2018 Feb;35(2):243-253. doi: 10.1007/s12325-017-0652-2. Epub 2017 Dec 21. PMID 29270781
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com